CLINICAL TRIAL: NCT06311123
Title: High Dimensional Mass Cytometry as a Tool to Understand Ozanimod's Mechanism of Action (MOA)
Brief Title: Understanding Ozanimod's MOA Via Mass Cytometry in Ulcerative Colitis
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: ISR IM047-059
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Chronic Moderate
Keywords: colitis; ozanimod; mass cytometry
MeSH Terms: conditions — Colitis, Ulcerative; Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with active ulcerative colitis: patients with active ulcerative colitis starting ozanimod therapy

SUMMARY:
The goal of this observational study is to learn about the mechanism of action of ozanimod in patients with ulcerative colitis (UC). The main questions it aims to answer are:

1. Prospectively assess the effects of ozanimod on the cellular composition of intestinal lamina propria and blood by deep immunophenotyping (CyTOF) of immune cell subsets prior and after the drug's administration.
2. Determine whether changes in cell subsets observed via mass cytometry correlate with with clinical or histologic parameters of disease activity.

Colonic biopsies and peripheral blood samples will be collected from patients with UC before and after the onset of ozanimod.

Researchers will compare intestinal and peripheral leukocytes before and after the drug's administration.

DETAILED DESCRIPTION:
Study Design/Methodology:

Several gastroenterologists at our center have agreed to assist with biopsy collection at our hospitals: UCSD: Singh, Boland, Patel, VA: Rivera-Nieves). Dr. Brian Behm who cares for most IBD patients at the University of Virginia has also agreed to assist with biopsy/PBMC collection.

During two visits (T0, T24-32) we will collect biopsies, endoscopies, histology, fecal and blood samples (Table 1), prospectively from a total of 10 UC patients scheduled for colonoscopy (before therapy with ozanimod and at 24-32 weeks post-treatment). A sample size of 10 patients per condition should be sufficient to achieve significant differences using CITRUS, based on required sample size determinations (see below).

The effects of the drug on cellular subsets will be assessed by comparing the two-time points (24-32 weeks post therapy) with its pretreatment control (T0). We will additionally compare the mass cytometry results to clinical parameters that are collected at our IBD center during every visit (Table 1). The clinical samples and parameters from patients recruited at UVA will be sent de-identified through a secure mailbox managed by the UVA.

Sample collection, storage, testing and analyses

1. After IV placement for conscious sedation, 10 mL of blood will be drawn on EDTA-containing tubes and sent to the lab on ice for further processing. Specimen transport is provided by staff from UCSD Center for Translational Research (CTRI). Upon arrival to the wet lab blood is spun, plasma separated and leukocytes isolated by gradient centrifugation. Cryopreservation media is added to the leukocyte fraction. Plasma and leukocytes are stored at -80 C.
2. Standard biopsies will also be obtained from ileum (control effect of drug on uninvolved segment), as well as in involved and uninvolved colonic segments and suspended in complete media for cell isolation. Specimen transport is provided by staff from UCSD Center for Translational Research. Upon arrival to the wet lab, cryopreservation media is added to the biopsies and stored at -80 C.

We have found significant batch to batch variation during pilot studies , even controlled using veri-cells. For that reason all cell/tissue processing and acquisition on the cytometer will all be performed together, upon completion of collection.

No study specific visits will be conducted for IBD patients. All visits and sample acquisitions will be at standard of care visits. No specific treatment related research interventions will be performed on IBD patients for this study. We thus categorize the the study as non-interventional.

Data Analysis:

We have been analyzing CyTOF data now for several years as illustrated in the two published manuscripts by Tyler et al.. In addition we have worked with Amir El-Ad who runs the AstoLabe platform for high dimensional cytometery analyses. To examine differences in population abundance and specific cell marker expression, we have identified CITRUS as one of many appropriate algorithms to perform our analysis of IBD biopsies. CITRUS identifies clusters of phenotypically similar cells in an unsupervised manner, characterizes the behavior of identified clusters using biologically interpretable metrics, and leverages regularized supervised learning algorithms to identify subset clusters whose behavior is predictive of the samples endpoint. CITRUS strongly encourages the use of a minimum of 8 samples per group. Thus, for our current project, we will obtain a minimum of 10 samples for UC before and after ozanimod therapy. As per estimates, based on our preliminary data, this sample size will be sufficient to accurately identify even rare populations and to determine changes in abundance between cell subsets. It is sensitive enough to assess differential expression of any marker in a three-way analysis. Bioinformatics comparisons between the cell subsets present in ileum, colon and PBMC at times 0 and 24-32 weeks for each patient will be performed for the principal endpoint of assessing the effect of the drug on relevant cell subsets.

Most recently, all of our data is stored in the Omiq platform, which provides multiple algorithms for data analyses.

For the univariable association of continuous independent variables with response, either an unpaired t-test or a Wilcoxon two-sample test will be used, while for categorical variables Fisher's exact test will used. All comparisons will be two-sided and performed at the 0.05 level of significance. As these analyses are exploratory, no adjustment will be made for multiple comparisons.

Data Management Plan: All data will be stored on password-protected computers at UCSD. All hard files and raw data will be stored in locked cabinets on UCSD campus within the lab of Jesus Rivera-Nieves. Patients will be given study identifiers as part of the IBD Biobank and no personal identifiers will be used. The Data Management plan will follow that of the UCSD IBD Biobank which has been extensively reviewed by the IRB and Committee for Protection of Human Subjects at UCSD.

At the UVA, data will be collected by the local study coordinator and de-identified. All data will be sent electronically using a secure mailbox. This has been approved by the UVA IRB.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 or older.
2. Have had UC diagnosed at least 3 months prior to screening. The diagnosis must be confirmed by endoscopic and histologic evidence.
3. Have active UC confirmed on endoscopy.
4. Ability to provide written informed consent to IBD biobank (UCSD)
5. Patients with above criteria being considered for ozanimod therapy and will not be treated in conjunction with biologics.

Exclusion Criteria:

1. Have severe IBD as evidenced by:physician judgment that the patient is likely to require colectomy or ileostomy within 12 weeks of baseline
2. Current evidence of fulminant colitis, toxic megacolon or bowel perforation
3. Previous total colectomy
4. Platelet count<100,000/μL
5. Have positive stool culture for pathogens (O+P, bacteria) or positive test for C. difficile at screening. If C. difficile is positive, the patient may be treated and retested.
6. Prisoners or subjects involuntarily detained will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe ulcerative colitis starting ozanimod therapy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
difference in leukocyte subsets | 3 years
  difference in leukocyte subsets as determined by mass cytometry analyses

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other interested investigators after approval by BMS
Supporting Information: Study Protocol, ICF
Time Frame: 10/2023 through 09/2026
Access Criteria: Data will be posted at website
URL: http://rci.ucsd.edu